CLINICAL TRIAL: NCT04102579
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy, Safety, and Tolerability of Valbenazine for the Treatment of Chorea Associated With Huntington Disease
Brief Title: Efficacy, Safety, and Tolerability of Valbenazine for the Treatment of Chorea Associated With Huntington Disease
Acronym: KINECT-HD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Collaborators: Huntington Study Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NBI-98854-HD3005
Record Dates: First submitted 2019-09-23; First posted 2019-09-25 (Actual); Results first posted 2023-10-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-09

CONDITIONS: Chorea, Huntington
Keywords: Huntington's; Huntington; Chorea; Movement disorder; Valbenazine; HD; Tetrabenazine; VMAT2-Inhibitor
MeSH Terms: conditions — Huntington Disease; Chorea; Movement Disorders | interventions — valbenazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Valbenazine (Experimental): Capsule, administered orally once daily for 12 weeks.
  Interventions: Drug: Valbenazine
- Placebo (Placebo Comparator): Capsule, administered orally once daily for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Valbenazine — vesicular monoamine transporter 2 (VMAT2) inhibitor
  Other Names: NBI-98854
  Arms: Valbenazine
Drug: Placebo — non-active dosage form
  Arms: Placebo

SUMMARY:
This is a Phase 3, randomized, double-blind, placebo-controlled study to evaluate the efficacy, safety, and tolerability of valbenazine to treat chorea in participants with Huntington disease.

ELIGIBILITY:
Inclusion Criteria:

1. Have a clinical diagnosis of Huntington Disease (HD) with chorea
2. Be able to walk, with or without the assistance of a person or device
3. Participants of childbearing potential who do not practice total abstinence must agree to use hormonal or two forms of nonhormonal contraception (dual contraception) consistently while participating in the study until 30 days (females) or 90 days (males) after the last dose of the study drug
4. Be able to read and understand English

Exclusion Criteria:

1. Have a history of previously established therapy with a VMAT2 inhibitor, in the judgement of the investigator
2. Have difficulty swallowing
3. Are currently pregnant or breastfeeding
4. Have a known history of long QT syndrome, cardiac tachyarrhythmia, left bundle-branch block, atrioventricular block, uncontrolled bradyarrhythmia, or heart failure
5. Have an unstable or serious medical or psychiatric illness
6. Have a significant risk of suicidal behavior
7. Have a history of substance dependence or substance (drug) or alcohol abuse, within 1 year of screening
8. If taking antidepressant therapy, be on a stable regimen
9. Have received gene therapy at any time
10. Have received an investigational drug in a clinical study within 30 days of the baseline visit or plan to use such investigational drug (other than valbenazine) during the study
11. Have had a blood loss ≥550 milliliters (mL) or donated blood within 30 days before the baseline visit
12. Had a medically significant illness within 30 days before baseline, or any history of neuroleptic malignant syndrome

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Chief Medical Officer
Locations (43):
- United States (40):
  - Neurocrine Clinical Site, Birmingham, Alabama
  - Neurocrine Clinical Site, Little Rock, Arkansas
  - Neurocrine Clinical Site, La Jolla, California
  - Neurocrine Clinical Site, Sacramento, California
  - Neurocrine Clinical Site, Aurora, Colorado
  - Neurocrine Clinical Site, Englewood, Colorado
  - Neurocrine Clinical Site, Washington D.C., District of Columbia
  - Neurocrine Clinical Site, Gainesville, Florida
  - Neurocrine Clinical Site, Miami, Florida
  - Neurocrine Clinical Site, Atlanta, Georgia
  - Neurocrine Clinical Site, Chicago, Illinois
  - Neurocrine Clinical Site, Indianapolis, Indiana
  - Neurocrine Clinical Site, Iowa City, Iowa
  - Neurocrine Clinical Site, Kansas City, Kansas
  - Neurocrine Clinical Site, Wichita, Kansas
  - Neurocrine Clinical Site, Louisville, Kentucky
  - Neurocrine Clinical Site, New Orleans, Louisiana
  - Neurocrine Clinical Site, Boston, Massachusetts
  - Neurocrine Clinical Site, Charlestown, Massachusetts
  - Neurocrine Clinical Site, Ann Arbor, Michigan
  - Neurocrine Clinical Site, West Bloomfield, Michigan
  - Neurocrine Clinical Site, Omaha, Nebraska
  - Neurocrine Clinical Site, Rochester, New York
  - Neurocrine Clinical Site, Williamsville, New York
  - Neurocrine Clinical Site, Durham, North Carolina
  - Neurocrine Clinical Site, Fargo, North Dakota
  - Neurocrine Clinical Site, Cleveland, Ohio
  - Neurocrine Clinical Site, Columbus, Ohio
  - Neurocrine Clinical Site, Toledo, Ohio
  - Neurocrine Clinical Site, Pittsburgh, Pennsylvania
  - Neurocrine Clinical Site, Charleston, South Carolina
  - Neurocrine Clinical Site, Columbia, South Carolina
  - Neurocrine Clinical Site, Greenville, South Carolina
  - Neurocrine Clinical Site, Nashville, Tennessee
  - Neurocrine Clinical Site, Houston, Texas
  - Neurocrine Clinical Site, Salt Lake City, Utah
  - Neurocrine Clinical Site, Burlington, Vermont
  - Neurocrine Clinical Site, Charlottesville, Virginia
  - Neurocrine Clinical Site, Seattle, Washington
  - Neurocrine Clinical Site, Spokane, Washington
- Canada (3):
  - Neurocrine Clinical Site, Vancouver, British Columbia
  - Neurocrine Clinical Site, Ottawa, Ontario
  - Neurocrine Clinical Site, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Furr Stimming E, Claassen DO, Kayson E, Goldstein J, Mehanna R, Zhang H, Liang GS, Haubenberger D; Huntington Study Group KINECT-HD Collaborators. Safety and efficacy of valbenazine for the treatment of chorea associated with Huntington's disease (KINECT-HD): a phase 3, randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2023 Jun;22(6):494-504. doi: 10.1016/S1474-4422(23)00127-8. PMID 37210099
- [Derived] Rodrigues FB, Wild EJ. Huntington's Disease Clinical Trials Corner: April 2020. J Huntingtons Dis. 2020;9(2):185-197. doi: 10.3233/JHD-200002. PMID 32250312
- See also: Study website — http://www.kinect-hd.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Valbenazine | Placebo
Started | 64 | 64
Received at Least 1 Dose of Study Drug | 64 | 63
Completed | 57 | 54
Not Completed | 7 | 10
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Lost to Follow-up | 0 | 1
Not completed — Discontinued Due to COVID-19-related Study Pause | 3 | 4
Not completed — Other than Specified | 1 | 0
Not completed — Not Dosed with Study Drug | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Valbenazine | Placebo | Total
Number analyzed (Participants) | 64 | 63 | 127
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (10.1) | 53.6 (11.6) | 53.8 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 36 | 69
  Male | 31 | 27 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 8
  Not Hispanic or Latino | 59 | 60 | 119
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 60 | 62 | 122
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  Canada | 2 | 7 | 9
  United States | 62 | 56 | 118

OUTCOME MEASURES:

1. Primary Outcome: Change From Screening Period Baseline to Maintenance Period in the Unified Huntington's Disease Rating Scale (UHDRS) Total Maximal Chorea (TMC) Score.
Description: The TMC is part of the motor assessment of the UHDRS and measures chorea in 7 different body parts including the face, oral-buccal-lingual region, trunk and each limb independently. The TMC score is the sum of the individual scores and ranges from 0 to 28. A decrease in TMC scores indicates improvement in chorea symptoms.
Time Frame: Baseline (average of screening and Day -1), maintenance (average of Weeks 10 and 12)
Population: All participants who are randomly assigned to a treatment group and who had at least 1 evaluable TMC change from baseline score during the 12-week double-blind treatment period.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Valbenazine | Placebo
Number analyzed (Participants) | 64 | 61
units on a scale | -4.60 (0.43) | -1.44 (0.44)
Statistical Analysis 1: Comparison: Valbenazine vs Placebo; Results were analyzed using a mixed-effect model repeated measures (MMRM) analysis. The model included the screening period baseline TMC as a covariate, and treatment group, visit, treatment group-by-visit interaction, and baseline-by-visit interaction as fixed effects. Participant was included as a random effect; Test type: Other; p < 0.0001, MMRM — Statistical significance achieved if p-value <0.05; Least Squares (LS) Means Difference = -3.16, 95% CI 2-sided [-4.37 to -1.95], Standard Error of Mean 0.61 — LS Means Difference = Valbenazine - Placebo

2. Secondary Outcome: Percent of Clinical Global Impression of Change (CGI-C) Responders at Week 12
Description: The CGI-C is a 7-point scale that rates the overall global change in chorea symptoms since the initiation of study drug dosing, ranging from 1 (very much improved) to 7 (very much worse), as assessed by the investigator or qualified clinician designee.
  Participants whose CGI-C score was either a 1 (very much improved) or a 2 (much improved) were classified as responders.
Time Frame: Week 12
Population: All participants who were randomly assigned to a treatment group, and who had at least 1 evaluable TMC change from baseline score and observed data at Week 12.
Measure: Number; unit: percentage of responders
Arm/Group | Valbenazine | Placebo
Number analyzed (Participants) | 56 | 53
percentage of responders | 42.9 | 13.2
Statistical Analysis 1: Comparison: Valbenazine vs Placebo; Test type: Other; p = 0.0007, Fisher Exact — Statistical significance achieved if p-value <0.05; Percent Difference in Responders = 29.65, 95% CI 2-sided [10.77 to 45.37] — Percent Difference in Responders (%) = Valbenazine - Placebo

3. Secondary Outcome: Percent of Patient Global Impression of Change (PGI-C) Responders at Week 12
Description: The PGI-C is a 7-point scale that rates the overall global change in chorea symptoms since the initiation of study drug dosing, ranging from 1 (very much improved) to 7 (very much worse), as assessed by the participant.
  Participants whose PGI-C score was either a 1 (very much improved) or a 2 (much improved) were classified as responders.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: percentage of responders
Arm/Group | Valbenazine | Placebo
Number analyzed (Participants) | 55 | 53
percentage of responders | 52.7 | 26.4
Statistical Analysis 1: Comparison: Valbenazine vs Placebo; Test type: Other; p = 0.0062, Fisher Exact — Statistical significance achieved if p-value <0.05; Percent Difference in Responders = 26.31, 95% CI 2-sided [6.32 to 43.74] — Percent Difference in Responders (%) = Valbenazine - Placebo

4. Secondary Outcome: Change From Baseline to Week 12 in the Quality of Life in Neurological Disorders (Neuro-QoL) Upper Extremity Function T-Score
Description: The Neuro-QoL Upper Extremity Function Short Form consists of 8 questions about physical abilities, rated from 1 (unable to do) to 5 (without any difficulty). The Neuro-QoL scores were standardized as T-scores with a mean of 50 and standard deviation of 10. Scores below 50 indicated below average upper extremity function. The change from baseline to Week 12 in the Neuro-QoL Upper Extremity Function T-score are presented here. An increase in score indicates increased function.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Valbenazine | Placebo
Number analyzed (Participants) | 64 | 61
units on a scale | -1.58 (1.01) | -3.00 (1.04)
Statistical Analysis 1: Comparison: Valbenazine vs Placebo; LS mean was based on the MMRM model which included corresponding baseline value of the Neuro-QoL Upper Extremity Function T-score as a covariate; treatment group, visit, baseline-by-visit interaction, and treatment group-by-visit interaction as fixed effects; and participant as a random effect; Test type: Other; p = 0.3304, MMRM — Statistical significance achieved if p-value <0.05; LS Means Difference = 1.42, 95% CI 2-sided [-1.46 to 4.31], Standard Error of Mean 1.46 — LS Means Difference = Valbenazine - Placebo

5. Secondary Outcome: Change From Baseline to Week 12 in the Neuro-QoL Lower Extremity Function T-Score
Description: The Neuro-QoL Lower Extremity Function Short Form consists of 8 questions about physical abilities, rated from 1 (unable to do) to 5 (without any difficulty). The Neuro-QoL scores were standardized as T-scores with a mean of 50 and standard deviation of 10. Scores below 50 indicated below average upper extremity function. The change from baseline to Week 12 in the Neuro-QoL Upper Extremity Function T-score are presented here. An increase in score indicates better function.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Valbenazine | Placebo
Number analyzed (Participants) | 64 | 61
units on a scale | -0.27 (0.82) | 0.61 (0.84)

ADVERSE EVENTS:
Time Frame: Day 1 (after dosing) through Week 14
Description: All-cause mortality, serious adverse events, and other adverse events were assessed using the safety analysis population which included all participants who were randomly assigned to a treatment group, received at least 1 dose of study treatment, and had any postbaseline safety data. Treatment-emergent adverse events were those that occurred on or after first dose date of study treatment and up to 14 days after the last dose of study treatment.
Arm/Group | Valbenazine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/64 | 1/63
Serious Adverse Events (participants affected / at risk) | 1/64 | 2/63
Other Adverse Events (participants affected / at risk) | 35/64 | 17/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Valbenazine (N=64) | Placebo (N=63)
Psychotic disorder (Psychiatric disorders) | 0 | 1
Colon cancer (Cardiac disorders) | 0 | 1 — A serious adverse event of colon cancer in the placebo group resulted in death.
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Valbenazine (N=64) | Placebo (N=63)
Fatigue (General disorders) | 9 | 6
Fall (Injury, poisoning and procedural complications) | 8 | 8
Somnolence (Nervous system disorders) | 10 | 2
Akathisia (Nervous system disorders) | 4 | 3
Rash (Skin and subcutaneous tissue disorders) | 5 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 5 | 0 — Note: One additional participant in the valbenazine group had an event of urticaria that was coded under the system organ class of immune system disorders.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, the PI has the right to publish results provided such publication does not violate confidentiality or IP provisions within the contract with the Sponsor. Prior to submission for publication or presentation of results, the PI must provide the Sponsor time for review. The Sponsor can request the PI to withhold or remove information from all publications. For a multi-center study, any publication of results by the PI shall not be made before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2021-04-12): https://cdn.clinicaltrials.gov/large-docs/79/NCT04102579/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-19): https://cdn.clinicaltrials.gov/large-docs/79/NCT04102579/SAP_001.pdf